CLINICAL TRIAL: NCT05182151
Title: Effect of Istradefylline Treatment on Behavioral Measures of Apathy in Parkinson's Disease.
Status: Terminated | Type: Observational
Why Stopped: recruitment issues
Sponsor: Medical University of South Carolina (Other)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00108116
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Apathy; Parkinson Disease
Keywords: istradefylline
MeSH Terms: conditions — Lethargy; Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient: istradefylline 40mg daily over 12 week period
  Interventions: Drug: Istradefylline 40 mg

INTERVENTIONS:
Drug: Istradefylline 40 mg — adenosine A2A receptor antagonist

SUMMARY:
Apathy is defined as a lack of feeling, emotion, interest, or concern. Apathy also involves reduction or loss of motivation and goal-directed behavior. Clinically significant apathy, where meaningful activities are given up and quality of life is diminished, is common in people with Parkinson's disease (PD).

Many individuals with Parkinson's disease experiencing fluctuations in the severity of their movement problems and medication "off" time. "Off" time refers to periods of the day between doses of PD medication when your motor symptoms (e.g., tremor, stiffness, slowness, walking problems, etc.) are worse and interfere with your ability to complete tasks of daily living. The investigational drug, Istradefylline, is an FDA-approved medication to treat motor fluctuations and "off" time in PD.

The purpose of this study is to investigate whether people with Parkinson's disease (PD) who are treated with istradefylline (ISD) show improvements in motivation and apathy over a 12-week period. Specifically, we wish to see whether people with PD who are treated with ISD engage in more physical and recreational activities, such as hobbies and other interests.

DETAILED DESCRIPTION:
Apathy is a clinical syndrome characterized by lack of motivation, interest, engagement, and emotional reactivity for goal-directed behaviors (Starkstein et al., 2008). A common and troublesome symptom in Parkinson's disease (PD), apathy is associated with diminished quality of life for both the patient and care partner (Van Reekum, Stuss, & Ostrander, 2005; Barone et al., 2009). To the extent that apathy reduces engagement in physical and social activities, it may also result in more rapid disease progression and cognitive decline (e.g., Crotty & Schwarzchild, 2020). Addressing apathy is therefore a crucial component of treating PD. A recent open-label study demonstrated significant reduction in self-reported apathy with Istradefylline (ISD) in PD (Nagayama et al, 2019). This unsurprising result likely reflects contributions from known benefits of ISD with respect to daytime somnolence and improved motor functioning (Matsuura et al., 2017; Suzuki et al. 2017), as well as enhanced functioning of dopamine-mediated reward pathways. However, patients with PD advanced enough to warrant treatment with ISD may also have diminished insight and awareness, and therefore not be particularly reliable reporters (e.g., Orfei et al., 2018). It is also unknown whether and to what extent this is correlated with actual changes in behavior and caregiver burden.

The objective of this study is to determine whether treatment with ISD increases engagement in physical and other meaningful activities in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PD consistent with United Kingdom Brain Bank Criteria or the Movement Disorder Society Research Criteria for the Diagnosis of Parkinson's Disease, with bradykinesia and sequence effect being present, and prominent motor asymmetry (if no rest tremor).
2. Current treatment with levodopa.
3. Stable on levodopa and other study-approved medications for PD motor symptoms for at least four weeks prior to screening.
4. Clinically significant wearing-off / fluctuating symptomatology warranting treatment with ISD
5. Presence of apathy at baseline (LARS > -22)
6. Living with adult informant

Exclusion Criteria:

Current or prior treatment with istradefylline. 2. History of Deep Brain Stimulation (DBS) surgery, ablative surgery (e.g., pallidotomy, thalamotomy, focused ultrasound, etc.), Duopa pump implantation, or other invasive intervention for Parkinson's disease symptoms. 3. Injury or concomitant health condition at screening that would preclude engagement in light physical activity. 10 4. Prior history of cerebrovascular accident (e.g., stroke or aneurysm) or seizure disorder (other than febrile seizures during childhood). 5. Dementia (MoCA<22) 6. Psychotic symptoms that would raise concern for safe use of ISD, as indicated by domains A (delusions) and B (hallucinations) of the Neuropsychiatric Inventory (NPI), and defined as a score of ≥4 on either the A (frequency × severity) or B (frequency × severity) scales of the NPI. 7. Depressive mood symptoms at baseline likely to interfere with response to treatment (BDI-II>19) 8. Active suicidal ideation within 1 year prior to Screening Visit as determined by a positive response to Question 4 or 5 on the C-SSRS. 9. Diagnosis or treatment for any central nervous system disorder other than Parkinson's disease that could be expected in the eyes of the investigator to impact ability to participate in study. 10. Contraindications / conditions that would preclude safe dosing of 40mg ISD 11. Change in medications for mood or anxiety within 6 weeks of enrollment or anticipation of change in medications for mood or anxiety during the 8-week study period. 12. Moderate or severe hepatic impairment. 13. Current treatment with strong CYP3A4 inhibitors 14. Current treatment with strong CYP3A4 inducers 15. Pregnant women are not able to participate due to unknown safety risks associated with ISD

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with dopaminergic therapy for idiopathic Parkinson's disease who have clinically significant motor fluctuations or "off" time warranting adjuvant treatment with ISD.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity Scale for the Elderly (PASE) | 12 weeks
  telephone survey

SECONDARY OUTCOMES:
Engagement in Meaningful Activities Survey (EMAS) | 12 weeks
  telephone survey
Lille Apathy Rating Scale (LARS) | 12 weeks
  apathy scale
Apathy Evaluation Scale (AES) | 12 weeks
  patient and informant
Beck Depression Inventory (BDI-2) | 12 weeks
  Depression scale
Epworth Sleepiness Scale (ESS) | 12 weeks
  scale to assess sleepiness
Global Impression of Change | 12 weeks
  patient and informant
Unified Parkinson's Disease Rating Scale | 12 weeks
  motor symptom rating

CONTACTS AND LOCATIONS:
Overall Officials: Lilia Lovera, MD, Study Chair — Medical University of South Carolina
Locations (1):
- MUSC Movement Disorders Program, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
None shared outside investigator group